CLINICAL TRIAL: NCT02318420
Title: The PartoMa Project for Saving Lives at Birth - An Intervention Based Study to Strengthen the Quality of Monitoring, Action and Triage During Labour at an East African Referral Hospital
Brief Title: The PartoMa Project: For Improving Monitoring, Action and Triage During Labour
Acronym: PartoMa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ib Christian Bygbjerg (Other)
Collaborators: University of Copenhagen (Other); Rigshospitalet, Denmark (Other); Free University Medical Center (Other); Mnazi Mmoja Hospital (Unknown); Lundbeck Foundation (Other); Laerdal Foundation (Other)
Responsible Party: Sponsor-Investigator, Ib Christian Bygbjerg, Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R164-2013-16038
Record Dates: First submitted 2014-11-04; First posted 2014-12-17 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Obstetric Labor Complications; Stillbirth; Maternal Death
Keywords: Obstetrics; Partogram; ePartogram; eHealth; Low-income; Quality of care; Perinatal death; Maternal death; Cesarean section; Health information technology
MeSH Terms: conditions — Obstetric Labor Complications; Stillbirth; Maternal Death; Perinatal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Women in labour (Experimental): All women in labour during the study period (4 months baseline and the 9th-12th month of the intervention) will be included for this pre- vs. post-study of the PartoMa intervention.
  The following subgroups will be studied in-depth:
  1. All stillbirths
  2. All maternal deaths
  3. All women with severe hypertensive disorders
  4. A randomized selected group of women delivering a the study site, approximately 300-600 each year.
  Interventions: Other: The PartoMa intervention
- Health care providers (Experimental): All health care providers (physicians and nurse-midwives) working at the Department of Obstetrics during the study period will be invited to participate in knowledge tests of obstetric care and qualitative participant observations as well as in-depth interviews regarding quality of care. This is a part of evaluating the use and effectiveness of the PartoMa intervention.
  Interventions: Other: The PartoMa intervention

INTERVENTIONS:
Other: The PartoMa intervention — WHO partogram, locally developed and achievable labour management guidelines (PartoMa guidelines), continual in-house training

SUMMARY:
OVERALL OBJECTIVE In an East African referral hospital, to develop and analyze the effect of locally agreed and achievable guidelines and a continual in-house training program for strengthening partogram-based monitoring-to-action during labour.

INTERVENTION Paper partograms (WHO), locally developed labour management guidelines (the PartoMa guidelines) and continual in-house education.

OVERALL DESIGN A quasi-experimental pre-post-study (The PartoMa study).

SETTING Department of Obstetrics and Gynaecology, Mnazi Mmoja Hospital, Zanzibar.

POPULATION Labouring women delivering at the study site from October 2014 to January 2016 and their offspring, as well as health providers. Women and their offspring will be enrolled at/after unset of labour and followed until discharge.

ENDPOINTS The primary composite endpoint is stillbirths and birth asphyxia. For further description and secondary outcomes, please see below.

STUDY TIME Data collection from October 2014 to January 2016, supplemented by a post-exit collection of case file data from October 2016 - January 2017.

DETAILED DESCRIPTION:
SPECIFIC OBJECTIVES

I (a) To analyze in depth current quality of intrapartum care by a mixed methods approach, including exploration of underlying challenges in care delivery and an association between suboptimal labour care and perinatal mortality. (b) To conduct a criterion-based audit of stillbirths investigating direct and indirect causes and related maternal risks.

II. To develop locally achievable and agreed partogram-associated labour monitoring-to-action guidelines (the PartoMa guidelines) for strengthening the partogram use as a decision support tool, and study its acceptability by skilled birth attendants.

III. To implement the PartoMa guidelines and low cost, low dose, high frequency, in-house training for strengthening the use of the partogram as a decision support tool, and study the effect on knowledge, skills, quality of intrapartum care, record keeping, and perinatal outcome.

IV. To conduct a post-exit 2 years evaluation of use and effect of the PartoMa guidelines and recurring training.

V. To develop an electronic smartphone application (the PartoMa app), which includes the PartoMa guidelines.

VI. To estimate the cost-effectiveness of the interventions studied (specific objectives III-V).

SETTING

The East African Mnazi Mmoja Hospital (MMH) in Zanzibar is a governmental referral facility serving the population of Zanzibar. As East Africa in general, the Zanzibarian archipelago struggles with poverty and a resource constraint health system, and half of the population live below the basic needs poverty line.

At the facility's Department of Obstetrics and Gynecology, the yearly number of deliveries is approximately 12,000. Approximately 50 maternal deaths occur annually (420 deaths per 100 000 live births). While the facility-based neonatal death rate is unknown, our baseline study revealed a stillbirth rate of 59 per 1000 total births, of which approximately half were alive at the time of admission.

Prior to this study, maternal and perinatal death audits were not conducted routinely and little is known about direct and indirect causes for the perinatal deaths.

METHODS

This study presents a quality improvement process of intrapartum monitoring, action and triage. The overall study design is here presented in relation to the four specific objectives:

I. The intervention-based study is based on an in-depth baseline quality of care assessment, which includes criterion-based audit of intrapartum management in cases of stillbirths compared to cases with Apgar scores of 7-10, and qualitative exploration of contributing causes to substandard labour management (including participant observations and in depth interviews).

II. Together with local doctors and nurse-midwives, international evidence-based guidelines are adapted to be locally achievable (the PartoMa guidelines). Additionally, they are internationally peer-reviewed with the aim of representing best possible care with the limited resources available at the facility.

III. A concept for reoccurring in-house training in monitoring-to-action during labour is developed, based on the PartoMa guidelines and implemented together with the guidelines. This PartoMa intervention (guidelines and reoccurring in-house training) is evaluated by comparing clinical practice and birth outcome (please see the specific outcome measures below) in the baseline period (October 2014 - January 2015) with the 9th-12th month of the intervention (October 2015 - January 2016).

IV. After the first intervention year (February 2016), a local steering group takes over the continual implementation of the PartoMa guidelines. If the intervention is still running, clinical practice and birth outcome will be analysed during the 21st - 24th month of the intervention (October 2016 - January 2017) and compared with previous assessments.

V. If the PartoMa guidelines show to be accepted among birth attendants and effective in improving quality of care, an electronic smartphone application (the PartoMa app) will be developed, which includes the PartoMa guidelines.

VI. A cost-effectiveness analysis of the intervention steps is carried out.

ELIGIBILITY:
Inclusion Criteria:

* All women in labour delivering at the study site and their outcome, October 2014 - January 2015 and October 2015 - January 2016
* All health care providers at the department during the baseline and intervention period, October 2014 - January 2016

For the different substudies, sub-groups are selected (please see the secondary outcomes for a description).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3087 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Composite outcome of stillbirths and birth asphyxia | A comparison of the baseline (Oct. 14 - Jan. '15) with 9th-12th month of the intervention (Oct. '15 - Jan. '16).
  Stillbirths (=late foetal deaths >=1000g), subdivided into pre- and intra-hospital stillbirths (with/without positive foetal heart rate on admission). Birth asphyxia was defined as newborns with a 5-minutes Apgar score < 6.

SECONDARY OUTCOMES:
Maternal death | A comparison of the baseline (Oct. 14 - Jan. '15) with 9th-12th month of the intervention (Oct. '15 - Jan. '16).
  Deaths of women at the study site while pregnant or within 42 days postpartum, from any cause related to or aggravated by pregnancy or its management.
Cesarean sections and vacuum extractions | A comparison of the baseline (Oct. 14 - Jan. '15) with 9th-12th month of the intervention (Oct. '15 - Jan. '16).
Process indicators of quality of intrapartum labour care | A comparison of the baseline (Oct. 14 - Jan. '15) with 9th-12th month of the intervention (Oct. '15 - Jan. '16).
  This includes partogram use, timely surveillance (of foetal heart rate, labour progress, and maternal vital signs), and oxytocin use for labour augmentation. Management is compared to pre-selected audit criteria.
Health providers' perception of their work situation in the labour and delivery rooms | This is assessed at multiple time points throughout the study period and more in-depth after 2 years of the intervention.
  Participant observations and in-depth interviews.
The women's experience of care received during delivery. | This is assessed through community visits in January - March 2016.
  By focus group discussions.
HALE | This will be evaluated economically after finalizing the study period.
  Cost of healthy life years gained /1,000 population /year

CONTACTS AND LOCATIONS:
Overall Officials: Ib C Bygbjerg, Professor, Study Director — University of Copenhagen; Nanna Maaløe, MD, Principal Investigator — University of Copenhagen
Locations (1):
- Dept. Obstetrics and Gynaecology, Mnazi Mmoja Hospital, Zanzibar, Zanzibar, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maaloe N, Andersen CB, Housseine N, Meguid T, Bygbjerg IC, van Roosmalen J. Effect of locally tailored clinical guidelines on intrapartum management of severe hypertensive disorders at Zanzibar's tertiary hospital (the PartoMa study). Int J Gynaecol Obstet. 2019 Jan;144(1):27-36. doi: 10.1002/ijgo.12692. Epub 2018 Oct 26. PMID 30307609
- [Derived] Maaloe N, Housseine N, van Roosmalen J, Bygbjerg IC, Tersbol BP, Khamis RS, Nielsen BB, Meguid T. Labour management guidelines for a Tanzanian referral hospital: The participatory development process and birth attendants' perceptions. BMC Pregnancy Childbirth. 2017 Jun 7;17(1):175. doi: 10.1186/s12884-017-1360-2. PMID 28592237
- [Derived] Maaloe N, Housseine N, Bygbjerg IC, Meguid T, Khamis RS, Mohamed AG, Nielsen BB, van Roosmalen J. Stillbirths and quality of care during labour at the low resource referral hospital of Zanzibar: a case-control study. BMC Pregnancy Childbirth. 2016 Nov 10;16(1):351. doi: 10.1186/s12884-016-1142-2. PMID 27832753